CLINICAL TRIAL: NCT05370729
Title: Impact of Combining N-acetylcysteine Intravenous Infusion and Intralipid Emulsion Infusion Versus Intralipid Infusion Alone on Myocardial Injury in Aluminum Phosphide Toxicity
Brief Title: Impact of N-acetylcysteine Infusion and Intralipid Infusion on Myocardial Injury in Aluminum Phosphide Toxicity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Tassbeeh Kamal, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NACILEALP
Record Dates: First submitted 2022-03-21; First posted 2022-05-11 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Myocardial Injury
Keywords: Aluminum phosphide poisonings; Intralipid emulsion; N-acetylcystiene; Myocardial injury; Echocardiography
MeSH Terms: interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- N-acetyl cysteine (NAC) (Experimental): Conservative management + ILE infusion 10 ml/hr + N-acetyl cysteine (NAC) infusion 150 mg/kg body weight in 200 ml of 5% dextrose over 1 h, followed by 50 mg/kg body weight in 500 ml of 5% dextrose over 4 h, and then 100 mg/kg body weight in 1000 ml of 5% dextrose over 16 h.
  Interventions: Drug: N-acetyl cysteine
- Intra lipid emulsion (ILE) (No Intervention): Conservative management + ILE infusion 10 ml/hr + normal saline infusion

INTERVENTIONS:
Drug: N-acetyl cysteine — Intravenous infusion of NAC 150 mg/kg body weight in 200 ml of 5% dextrose over 1 h, followed by 50 mg/kg body weight in 500 ml of 5% dextrose over 4 h, and then 100 mg/kg body weight in 1000 ml of 5% dextrose over 16 h.
  Other Names: NAC
  Arms: N-acetyl cysteine (NAC)

SUMMARY:
Assess impact of ILE and NAC in morbidity and mortality when used as adjuvant therapy to routine management of acute ALP poisoning.

DETAILED DESCRIPTION:
Aluminum phosphide (ALP) is one of the solid fumigant pesticides. In Egypt, ALP is extensively used to protect grains against insects and rodents. It is available in the form of tablets known as "grain tablet". Suicidal ingestion of ALP tablets is obviously increasing in developing countries. This is attributed to its wide use, free availability in the market, and its low cost.

Aluminum phosphide toxicity is extremely fatal. The conveyed mortality rate differs from 37-100%. More than 90% of patients die within the first 24 hours, mainly due to cardiac dysrhythmia. Despite continuous research, no effective antidote has been reported for this lethal poisoning so far. PH3 is phosphorus trihydride and solubility of phosphorus can affect PH3. Solubilities of phosphorus are as follows: In water: 1 part/300,000 parts water; in absolute alcohol: 1 g/400 mL. One gram phosphorus dissolves in 80 ml olive oil, 60 ml oil of turpentine, and about 100 mL of almond oil. So, PH3 might also have lipid soluble property and used IV lipid emulsion may counter its effects.

Intravenous lipid emulsion (ILE) is a sterile fat emulsion prepared for intravenous administration as a source of calories and essential fatty acids. Its main components include up to 20% soybean oil, 1.2% egg yolk phospholipids, 2.25% glycerin, and water for injection. In addition, sodium hydroxide has been added to adjust the pH, so that the final pH is 8.

Based on animal models and clinical studies, ILE is an established antidote for local-anesthetic drugs systemic toxicity. Besides, ILE has been well used for resuscitation of severe toxicities caused by various lipophilic non-local anesthetic drugs.

N-acetylcysteine (NAC) is a well-studied compound which is commonly used in the treatment of paracetamol poisoning. It has shown to replenish cellular glutathione stores in addition to the strong antioxidant properties. NAC has shown to reduce mortality, hospitalization time, and need for mechanical ventilation in ALP poisoning. A cohort study by Agarwal reported survival benefit in patients who received treatment with NAC compared to the control group.

Brain natriuretic peptide (BNP) is an excellent biomarker because it can be detected in the early stages of ischemia and decreases shortly after ischemia allowing better detection of re-injury. A metabolite of BNP, Nterminal pro-BNP, NT-proBNP, is relatively easy to measure and predicts short and long term outcomes. BNP is a 32-amino-acid peptide synthesized predominantly from the ventricular myocardium and is released in proportion to the degree of wall stress. Although it has gained recent prominence in the diagnosis and treatment of heart failure, BNP has recently shown promise in predicting the extent of myocardial ischemia in acute coronary syndromes. For instance, the magnitude of BNP released between 1 and 7 days after a myocardial infarction is predictive of left ventricular dysfunction, heart failure, and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Presentation with symptomatic acute ALP poisoning.
* History of exposure including reliable identification of the compound based on the container brought by patient's relatives.
* The suggestive clinical manifestations following shortly after a single exposure to ALP.

Exclusion Criteria:

* Co-ingestion or exposure to other substances in addition to ALP.
* Patients had major medical conditions (e.g., cardiovascular disease, renal or hepatic failure).
* Patients received treatment in any hospital or medical center before admission - other than emergency department of Assiut University Hospital.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Echocardiography | 24 hours
  Follow up cardiac function by echocardiography focusing on LV EF

SECONDARY OUTCOMES:
Renal function test | 24 hours
  Effect on renal function by measuring serum creatinine and serum BUN
Total days of ICU stay | Up to two weeks
  ICU stay

CONTACTS AND LOCATIONS:
Overall Officials: Ola M Wahba, PHD, MD, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baruah U, Sahni A, Sachdeva HC. Successful management of aluminium phosphide poisoning using intravenous lipid emulsion: Report of two cases. Indian J Crit Care Med. 2015 Dec;19(12):735-8. doi: 10.4103/0972-5229.171412. PMID 26816450
- [Background] Tehrani H, Halvaie Z, Shadnia S, Soltaninejad K, Abdollahi M. Protective effects of N-acetylcysteine on aluminum phosphide-induced oxidative stress in acute human poisoning. Clin Toxicol (Phila). 2013 Jan;51(1):23-8. doi: 10.3109/15563650.2012.743029. Epub 2012 Nov 14. PMID 23148565
- [Background] Agarwal A, Robo R, Jain N, Gutch M, Consil S, Kumar S. Oxidative stress determined through the levels of antioxidant enzymes and the effect of N-acetylcysteine in aluminum phosphide poisoning. Indian J Crit Care Med. 2014 Oct;18(10):666-71. doi: 10.4103/0972-5229.142176. PMID 25316977
- [Background] Tsutamoto T, Wada A, Maeda K, Hisanaga T, Maeda Y, Fukai D, Ohnishi M, Sugimoto Y, Kinoshita M. Attenuation of compensation of endogenous cardiac natriuretic peptide system in chronic heart failure: prognostic role of plasma brain natriuretic peptide concentration in patients with chronic symptomatic left ventricular dysfunction. Circulation. 1997 Jul 15;96(2):509-16. doi: 10.1161/01.cir.96.2.509. PMID 9244219